CLINICAL TRIAL: NCT00177125
Title: Evaluating the Effect of the Vacuum Constriction Device on Erectile Function and Penile Length Post Radical Retropubic Prostatectomy
Brief Title: Evaluating the Effect of the VCD on Erectile Function and Penile Length Post RRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Endocare, Inc. (Industry); Manoj, Monga, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0406M61241; 3358B
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Prostatic Neoplasms; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ErectAid

SUMMARY:
The purpose of this study is to perform a randomized prospective study to evaluate whether the vacuum erection device facilitates an earlier return of erectile function post radical prostatectomy. A secondary measure will be to evaluate if the vacuum erection device can help prevent penile shortening.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a radical prostatectomy for prostate cancer who are able to attain a partial or full erection preoperatively and are sexually active.

Exclusion Criteria:

* Patients on anticoagulation therapy and those with bleeding diatheses
* Insufficient manual dexterity of patient or spouse
* IIEF(International Index of Erectile Function) at baseline < 11, indicating severe erectile dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2004-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, MD, Principal Investigator — University of Minnesota and VAMC Minneapolis
Locations (2):
- United States (2):
  - VAMC Minneapolis, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota